CLINICAL TRIAL: NCT01406340
Title: A Repeat-dose, Open-label, Parallel-group Study to Assess the Pharmacokinetics of GSK1278863 and Metabolites in Normal Subjects and Subjects With Impaired Renal Function
Brief Title: Assessment of the Pharmacokinetics of GSK1278863 and Metabolites in Normal Subjects and Subjects With Renal Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty enrolling last cohort of subjects
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 115573
Record Dates: First submitted 2011-07-26; First posted 2011-08-01 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Anaemia
MeSH Terms: conditions — Anemia | interventions — GSK1278863

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal subjects and subjects with Stage 3/4 renal function (Experimental): Subjects will receive 5mg GSK1278863 for 14 days.
  Interventions: Drug: 5 mg GSK1278863
- Subjects with Stage 5 renal function (Experimental): Subjects will receive 5mg GSK1278863 for 15 days.
  Interventions: Drug: 5 mg GSK1278863

INTERVENTIONS:
Drug: 5 mg GSK1278863 — 5 mg per day administered orally for 14 days for normal subjects and subjects with Stage 3/4 renal function; 5 mg per day administered orally for 15 days for subjects with Stage 5 renal function

SUMMARY:
This will be an open-label, parallel-group study to evaluate the pharmacokinetics of GSK1278863 and metabolites in normal subjects and subjects with impaired renal function, including those who are hemodialysis dependent. GSK1278863 will be administered once daily for 14 days to normal subjects and subjects with Stage 3 and Stage 4 renal function, and 15 days to subjects with Stage 5 renal function. Pharmacokinetic assessments will be made on Days 1 and 14 (normal subjects, subjects with Stage 3 and Stage 4 renal function) or Days 14 and 15 (dialysis and non-dialysis days; Stage 5).

ELIGIBILITY:
Inclusion Criteria:

All Study Participants

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Adults between 18 and 75 years of age at the time of Screening.
* A female subject is eligible to participate if she is of childbearing potential, and must agree to use one of the contraception methods described in the protocol. This criterion must be followed from the time of Screening until completion of the Follow-up Visit. OR Non-childbearing potential as defined in the protocol.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods in the protocol. This criterion must be followed from the time of the first dose of investigational product until completion of the Follow-up visit.
* Satisfactory medical evaluation based upon medical history, medication history, physical examination, and clinical laboratory data obtained at the screening visit.
* Body weight ≥ 45 kg and ≤ 140 kg at screening. For Stage 5 subjects, body weight is dry weight after hemodialysis.
* QTcF < 450 msec; OR QTcF < 480 msec in subjects with Bundle Branch Block. These should be based on average of triplicate values obtained over brief recording period at screening and Predose on Day 1.
* Vitamin B12 and folate above the lower limit of normal at screening.
* The subject is mentally and legally able to comply with the requirements and restrictions of the protocol and has provided signed informed consent prior to participation in any protocol-specific procedures, including screening procedures.

Additional Inclusion Criteria for Subjects with Normal Renal Function

* Has normal creatinine clearance (CLCR) via the Cockcroft-Gault equation, using serum creatinine and demographic data, obtained at Screening. Normal subjects should have no greater than trace blood or protein on Screening urinalysis.
* A hemoglobin value at screening is greater than the lower limit of the reference range for the local laboratory and less than or equal to 16.0g/dL
* No greater than trace blood on screening urinalysis
* Laboratory values for which specific criteria are not defined within the inclusion and exclusion criteria for this study must be within the normal range or deemed not clinically significant. A normal subject with a clinical abnormality or laboratory parameters outside the reference range may be included only if the investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures, or the integrity of the study.

Additional Inclusion Criteria for Subjects with Renal Impairment

* Has Stage 3 or Stage 4 renal function (not receiving dialysis) as determined by estimated Glomerular Filtration Rate (eGFR) calculated by the abbreviated MDRD equation OR has Stage 5 renal function (end-stage renal failure) and has been on stable hemodialysis treatment scheduled three times weekly for 3 months prior to screening and the serum creatinine value at the Day -1 visit must be within +/- 20% of the screening value.
* Is otherwise considered clinically stable with respect to underlying renal impairment as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG.
* has clinical laboratory test results that are considered clinically stable in the opinion of the Investigator, especially if the clinical abnormality or laboratory parameter is deemed associated with the subject's underlying renal impairment.
* has AST, ALT, alkaline phosphatase and bilirubin < or = 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Meets the following erythropoiesis stimulating agent (ESA) criteria: The subject is ESA naïve OR the subject has a scheduled ESA interval which is ≤ 7 days, ESA treatment must be discontinued for at least 7 days OR the subject has a scheduled ESA interval which is > 7 days, ESA treatment must be discontinued for at least that scheduled interval length (e.g. discontinued ≥ 14 days for a scheduled 14 day ESA interval) AND the subject will not resume ESA treatment until completion of the Follow-up Visit.
* Has a hemoglobin value: For ESA naïve subjects: ≤11.0 g/dL or subjects receiving ongoing ESA treatment: ≤12.0 g/dL at screening with a re check value of ≤11.0 g/dL after appropriate ESA discontinuation according to the Inclusion criterion on use of ESAs and prior to commencing investigational product dosing.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

All Study Participants

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result at Screening.
* A positive test for HIV antibody.
* Uncontrolled hypertension (diastolic BP >100 mmHg or systolic BP >160 mmHg at Screening.
* A positive drugs of abuse and alcohol screen.
* History of regular alcohol consumption within 6 months of the study as described in the protocol.
* History of regular use of tobacco- or nicotine-containing products within 6 months of the study in excess of 20 cigarettes per day or equivalent.
* History of drug abuse or dependence within 6 months of the study.
* History of sensitivity to any of the investigational products, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* The subject has participated in a clinical trial and has received an experimental investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if the clinical research unit uses heparin to maintain intravenous cannula patency).
* History of thrombosis defined as deep vein thrombosis, stroke, pulmonary embolism or other thrombosis related condition within 1 year prior to Screening.
* History of myocardial infarction or acute coronary syndrome within 1 year prior to Screening
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, and/or hepatic function that could interfere with the absorption, metabolism, and/or excretion of the investigational product. Examples of conditions that could interfere with normal gastrointestinal anatomy or motility include cholecystectomy, gastrointestinal bypass surgery, partial or total gastrectomy, small bowel resection, vagotomy, malabsorption, Crohn's disease, ulcerative colitis, or celiac sprue. Examples of conditions that could interfere with hepatic function include Gilbert's syndrome.
* Evidence of active peptic, duodenal or esophageal ulcer disease at Screening.
* History of chronic rectal bleeding.
* Subjects with polycystic kidney disease.
* Subjects with chronic inflammatory disease that could impact erythropoiesis (e.g., scleroderma, systemic lupus erythematosis, rheumatoid arthritis, celiac disease).
* Subjects with chronic lung disease requiring supplemental oxygen.
* Patients with a diagnosis of pulmonary artery hypertension.
* Subjects with Class III or Class IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system.
* Post-renal transplantation subjects with functioning transplant. Note: Failed transplant subjects back on hemodialysis are eligible for participating in this study but should not be on immunosuppressive medications for past 3 months at Screening.
* Active malignancy or diagnosis of malignancy within 5 years prior to screening (excluding successfully treated basal or squamous cell carcinoma).
* History of proliferative vascular eye disease (e.g., choroidal or retinal disease, such as neovascular age-related macular degeneration or proliferative diabetic retinopathy or wet macular edema) based on verbal confirmation having had an ophthalmologic exam within 12 months of screening.
* Pregnant females as determined by positive serum beta-hCG test at Screening and Day -1.
* Lactating females.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures, or lifestyle and/or dietary restrictions outlined in the informed consent and as directed by site staff.
* Consumption of red wine, grapefruit (juice), blood orange (juice), star fruit, onions, kale, broccoli, green beans, or apples from 7 days prior to the first dose of investigational product, unless in the opinion of the Investigator and GSK Medical Monitor this will not interfere with the study procedures and compromise subject safety.
* Subject is either an immediate family member of a participating investigator, study coordinator, employee of an investigator; or is a member of the staff conducting the study.

Additional Exclusion Criteria for Subjects with Normal Renal Function

* The values of hematological parameters at screening are outside the reference range and deemed clinically significant by the Investigator or GSK Medical Monitor.
* The values of the following tests at screening are: - TIBC: outside the reference range and serum iron: outside the reference range and serum ferritin: outside the reference range.
* Use or planned use of any prescription or non-prescription drugs that are prohibited as defined in the protocol within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of investigational product until completion of the follow-up visit unless in the opinion of the investigator or GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.

Additional Exclusion Criteria for Subjects with Renal Impairment

* The values of ferritin and transferrin at Screening for renal impaired subjects are: transferrin saturation ≥ 20% and serum ferritin < 100 μg/L
* Taking a prohibited medication or supplement (with the exception of approved vitamins or minerals within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of investigational product until completion of the follow-up visit, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study. The following medications are specifically prohibited from screening to the follow-up visit: non-steroidal anti-inflammatory drugs (NSAID) and immunosuppressant drugs and drugs used to treat malignancies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-08-30 (Actual); Primary Completion 2013-08-31 (Actual); Study Completion 2013-08-31 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve over the dosing interval . Composite of Pharmacokinetics | Blood samples will be collected at predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 and 72hr post dosing on Day 1 and Day 14 for normal and Stage3/4 subjects, and on Day 14 and Day 15 for Stage 5 subjects
  Area under the concentration-time curve over the dosing interval of GSK1278863 and metabolites on Day 1 and Day 14 for normal subjects and subjects with Stage 3/4 renal function; Area under the concentration-time curve over the dosing interval of GSK1278863 and metabolites on Day 14 (dialysis) and Day 15 (non-dialysis) for subjects with Stage 5 renal function.
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time. Composite of Pharmacokinetics | Blood samples will be collected at predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 and 72hr post dosing on Day 1 in normal and Stage3/4 subjects
  Area under the concentration-time curve from time zero (pre-dose) of GSK1278863 and metabolites on Day 1 for normal subjects and subjects with Stage 3/4 renal functione-dose) extrapolated to infinite time for
Maximum observed concentration. Composite of Pharmacokinetics | Blood samples will be collected at predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 and 72hr post dosing on Day 1 and Day 14 for normal and Stage3/4 subjects, and on Day 14 and Day 15 for Stage 5 subjects
  Maximum observed concentration of GSK1278863 and metabolites on Day 1 and Day 14 for normal subjects and subjects with Stage 3/4 renal function; Maximum observed concentration of GSK1278863 and metabolites on Day 14 and Day 15 for subjects with Stage 5 renal function.

SECONDARY OUTCOMES:
Safety and tolerability as assessed by the number of adverse events during the dosing period. | For normal subjects and subjects with Stage 3/4 renal function, from Day 1 to the follow-up visit at approximately Day 27. For subjects with Stage 5 renal function, from Day 1 to the follow-up visit at approximately Day 28.
Time of occurrence of maximum observed concentration | Day 1 and Day 14
  Time of occurrence of maximum observed concentration of GSK1278863 and metabolites on Day 1 and Day 14 for normal subjects and subjects with Stage 3/4 renal function
Terminal phase half-life | Day 1 and Day 14
  Terminal phase half-life of GSK1278863 and metabolites on Day 1 and Day 14 for normal subjects and subjects with Stage 3/4 renal function
renal clearance | Day 14
  renal clearance of GSK1278863 and metabolites in normal subjects and subjects with Stage 3/4 renal function
dialysis clearance | Day 14
  dialysis clearance of GSK1278863 and metabolites in Stage 5 renal function
change from baseline in QTcB or QTcF | For normal subjects and subjects with Stage 3/4 renal function, from Day 1 to Day 14; For subjects with Stage 5 renal function, from day 1 to day 15.
change from baseline in heart rate | For normal subjects and subjects with Stage 3/4 renal function, from Day 1 to the follow-up visit at approximately Day 27. For subjects with Stage 5 renal function, from Day 1 to the follow-up visit at approximately Day 28.
Safety and tolerability of GSK1278863 as assessed by change from baseline in toxicity grading of clinical laboratory tests | For normal subjects and subjects with Stage 3/4 renal function, from Day 1 to Day 15; For subjects with Stage 5 renal function, from Day 1 to Day 16.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=200942

REFERENCES:
- [Background] Caltabiano S, Cizman B, Burns O, Mahar KM, Johnson BM, Ramanjineyulu B, Serbest G, Cobitz AR. Effect of renal function and dialysis modality on daprodustat and predominant metabolite exposure. Clin Kidney J. 2019 Feb 18;12(5):693-701. doi: 10.1093/ckj/sfz013. eCollection 2019 Oct. PMID 31583094
- See also: Results for study 115573 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115573?search=study&search_terms=115573#rs